CLINICAL TRIAL: NCT06287892
Title: Diagnosis of Hypertrophic Cardiomyopathy With Artificial Intelligence-enhanced Electrocardiogram
Brief Title: Diagnosis of HCM With AI-ECG
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Yixiu Liang, Director of Department of Cardiology, Shanghai Zhongshan Hospital
Other Study IDs: AI-ECG-HCM
Record Dates: First submitted 2023-04-08; First posted 2024-03-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCM group: Patients diagnosed with HCM
- Control group: Subjects without HCM

SUMMARY:
The study aims to establish a diagnostic model of hypertrophic cardiomyopathy with artificial intelligence-enhanced electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCM

Exclusion Criteria:

* Patients with ventricular pacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes patients with HCM, and subjects without HCM as control.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of HCM with AI-ECG | 1 year within the time frame of ECG data collection
  First a diagnosis of HCM is made as the standard outcome according to 1) an International Classification of Diseases (ICD) code for HCM (ICD-9425.1, 425.11, 425.18, and ICD10 I42.1, I42.2); 2) reports from the echocardiographers.
  An AI-ECG algorithm will be used to make a diagnosis of HCM and compared with the standard outcome.
  The performance of the AI-ECG algorithm will be evaluated with metrics including AU-ROC, specificity, sensitivity and F1 value.

CONTACTS AND LOCATIONS:
Overall Officials: Yixiu Liang, MD, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No